CLINICAL TRIAL: NCT06636929
Title: Effect of Problematic Smartphone Use on Upper Extremity Functions and Cognitive Functions
Brief Title: Effect of Problematic Smartphone Use
Status: Active, not recruiting | Type: Observational
Sponsor: Kutahya Health Sciences University (Other)
Responsible Party: Principal Investigator, Ismail Okur, Assist. Prof., Kutahya Health Sciences University
Other Study IDs: KSBU 2024/04-27
Record Dates: First submitted 2024-10-08; First posted 2024-10-15 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Smartphone Addiction
Keywords: problematic smartphone use; smartphone addiction; cognitive function; reaction time; upper extremity problem
MeSH Terms: conditions — Internet Addiction Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: Participants with problematic smartphone use were identified with the Smartphone Addiction Scale Short Form. Participants with a score above 31 for women and 33 for men were defined as individuals with problematic smartphone use.
- Control group: Participants with problematic smartphone use were identified with the Smartphone Addiction Scale Short Form. Participants with a score below 31 for women and 33 for men were defined as the control group.

SUMMARY:
There is no study that examines the effect of problematic use of smartphones, which has become a global problem today, on reaction time and cognitive functions together. This study was planned to examine the effect of problematic smartphone use on upper extremity functions and cognitive functions. Participants' problematic smartphone use will be evaluated with the Smartphone Addiction Scale Short Form. Within the scope of upper extremity functions, Quick Disabilities of Arm, Shoulder & Hand Questionnaire, reaction time and grip strength will be evaluated. Reaction time will be measured with BlazePod Trainer (Blazepod Trainer Device, Play Coyotta Ltd, Tel Aviv, Israel). Jamar dynamometer (Performance Health, Warrenville, IL) will be used to evaluate grip strength. Cognitive functions will be assessed using the Stroop Test ÇAPA Form, Trail Making Test and Cognitive Failures Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* To be between 18-25 years old
* Using a smartphone for at least 1 hour a day
* Volunteering to participate in the study

Exclusion Criteria:

* Having undergone a surgical operation involving the upper extremity within the last 6 months
* History of trauma to the shoulder, elbow, hand and wrist in the last 6 months
* Presence of a diagnosed neurological, rheumatic or psychiatric disease

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adults aged 18-25 years
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2024-10-20 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Smartphone Addiction Scale Short Form | Baseline
  It is a 10-item scale to assess problematic smartphone use. Each item in the scale is scored between 1 (strongly disagree) and 6 (strongly agree). The total score ranges from 10-60, with higher scores indicating an increased risk of smartphone addiction. The cut-off score of the scale was reported as 33 for women and 31 for men.
Upper Extremity Functions-Quick Disabilities of Arm, Shoulder & Hand (Quick DASH) | Baseline
  In the 11-question scale, difficulties encountered during activities of daily living (carrying shopping bags, opening jars, using a knife to cut food, etc.) due to problems in the shoulder, elbow and hand regions are scored from 1 (no difficulty) to 5 (no difficulty at all). A higher total score indicates an increased level of functional limitation in the upper limb.
Upper Extremity Functions-Reaction Time | Baseline
  The upper extremity reaction time will be assessed using the BlazePod Trainer (Blazepod Trainer Device, Play Coyotta Ltd, Tel Aviv, Israel). Participants will be asked to hit 5 LEDs on a table as quickly as possible using only one hand while in a seated position. The LEDs will be arranged in an arc on the table within the participant's reach without disturbing their seated posture. The right and left hands will be evaluated separately. The number of LEDs hit in 30 seconds, the unit hit time (ms), and the number of missed LEDs (those that automatically hit after a 5-second waiting period) will be recorded through the BlazePod app installed on the researchers' phones.
Upper Extremity Functions-Grip Strength | Baseline
  A calibrated digital Jamar dynamometer (Performance Health, Warrenville, IL) will be used for grip strength. Participants will be instructed to squeeze the dynamometer as hard as possible while sitting in an upright position as recommended by the American Society of Hand Therapists, with arms at their sides, elbows flexed 90° and forearms in a neutral position. For hand grip strength, 3 measurements will be made with one minute intervals between each measurement and the average value will be recorded.
Cognitive Functions-Stroop Test ÇAPA Form | Baseline
  It is used to assess executive functions such as attention, information processing speed and response inhibition. The Stroop Test ÇAPA Form consists of a total of 60 items. In the first part, there are small rectangles (0.5 x 1 cm) with colors such as yellow, blue and red. In the second part, there are color names written in different colors. The test is administered in 3 stages. In the first part (Stroop A), the person is asked to name the colors in the boxes from left to right. If a color blindness is detected, the test can be terminated. In the second part (Stroop B), the person is asked to read quickly the color names written in different colors (yellow, red, green). In the third part (Stroop C), participants are asked to say the colors of the words (blue, green, yellow) without reading the color names. In all three parts, the time is timed and recorded with a stopwatch.
Cognitive Functions-Trail Making Test | Baseline
  It is used to assess cognitive functions such as working memory, complex attention and cognitive flexibility. It requires visual scanning and hand-eye coordination. The Trail Making Test consists of 25 circles with numbers distributed on paper and has 2 sections (IST A-B). Section A contains numbers numbered between 1 and 25, and during the test, individuals are asked to connect the circles by drawing lines consecutively and in the correct order. In part B, the circles contain both numbers and letters. Participants are asked to quickly connect the circles in consecutive order in accordance with the order of numbers and letters (1-A, 2-B, 3-C, etc.) by drawing a line without lifting the pencil from the paper. The time to complete each trace is recorded in seconds (s), A and B.
Cognitive Functions-Cognitive Failures Questionnaire | Baseline
  Errors in perception, memory and motor functions in daily life are assessed with 25 questions. Each question is scored from 0 (never) to 4 (very often). The total score ranges from 0-100, with a higher score indicating an increased level of cognitive error.

CONTACTS AND LOCATIONS:
Overall Officials: Ismail Okur, PT, PhD, Principal Investigator — Kutahya Health Sciences University
Locations (1):
- Kutahya Health Sciences University, Kütahya, Center, Turkey (Türkiye)